CLINICAL TRIAL: NCT02368379
Title: Diagnosis of Central Adrenal Insufficiency in Patients With Prader-Willi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Manmohan Kamboj, Associate Professor of Pediatrics, Section of Endocrinology, Metabolism and Diabetes, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 293113
Record Dates: First submitted 2015-02-05; First posted 2015-02-23 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Prader Willi Syndrome; Adrenal Insufficiency
Keywords: Metyrapone; ACTH stimulation test
MeSH Terms: conditions — Prader-Willi Syndrome; Adrenal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assessment of Central Adrenal Insufficiency (Other): Patients will undergo low dose ACTH stimulation test followed by overnight metyrapone test to assess for central adrenal insufficiency.
  Interventions: Other: Low dose (1 mcg) ACTH stimulation test; Other: Overnight metyrapone test

INTERVENTIONS:
Other: Low dose (1 mcg) ACTH stimulation test — Subjects will have baseline cortisol and ACTH drawn followed by administration of 1 mcg/m2 (max 1 mcg) of cortrosyn. Blood will be drawn at 20 and 40 minutes post cortrosyn for peak cortisol assessment of central adrenal insufficiency.
Other: Overnight metyrapone test — Subjects will receive metyrapone 30 mg/kg (max 3 grams) by mouth at midnight. Blood will be drawn at 0800 AM the following morning for ACTH, cortisol and 11 deoxycortisol for assessment of central adrenal insufficiency.

SUMMARY:
The purpose of this study is to determine presence of central adrenal insufficiency in children with Prader Willi Syndrome using low dose (1 mcg) ACTH stimulation test compared to results of overnight metyrapone test.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Prader Willi Syndrome ages 2 years and older

Exclusion Criteria:

* Individuals who are ill at the time of study
* Individuals who are pregnant at the time of study
* Individuals who it is deemed unsafe to stop taking medications known to affect the results of they study (hydrocortisone, phenytoin, estrogen, acetaminophen, oral anti-diabetic agents).

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Presence of central adrenal insufficiency using low dose (1 mcg) ACTH stimulation test | 40 minutes
Prescence of central adrenal insufficiency using overnight metyrapone test | 8 hours

SECONDARY OUTCOMES:
Determine peak cortisol value on low dose (1 mcg) ACTH stimulation test that can accurately predict central adrenal insufficiency based on overnight metyrapone test with good sensitivity and specificity. | 0

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States